# APPENDIX A – ACTIV-5/BET-A: RISANKIZUMAB/REMDESIVIR VS. PLACEBO/REMDESIVIR

## **TABLE OF CONTENTS**

| Appendix A – ACTIV-5/BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir | I |
|---|---|
| TABLE OF CONTENTS | 2 |
| LIST OF TABLES | 3 |
| 1. PROTOCOL SUMMARY | |
| 1.1 Synopsis | |
| 1.2 Schedule of Assessments | |
| 2. INTRODUCTION | 7 |
| 2.1 Study Rationale | - |
| 2.2 Background | |
| 2.2.1 Purpose of Study | |
| 2.2.2 Potential Therapeutic Agents | |
| 2.3 Risk/Benefit Assessment | |
| 2.3.2 Potential Risks of Remdesivir | |
| 2.3.3 Potential Risks of Risankizumab | |
| 2.3.4 Known Potential Benefits | |
| 3. OBJECTIVES AND ENDPOINTS | 10 |
| 4. STUDY DESIGN | 14 |
| 4.1 Overall Design | |
| 4.2 Justification for Dose | |
| <ul><li>4.2.1 Justification for Dose of Remdesivir</li></ul> | |
| 5. STUDY POPULATION | |
| <ul><li>5.1 Inclusion Criteria</li><li>5.2 Exclusion Criteria</li></ul> | |
| 5.2.1 Exclusion of Specific Populations | |
| 5.3 Inclusion of Vulnerable Subjects | |
| <ul><li>5.4 Lifestyle Considerations</li><li>5.5 Screen Failures</li></ul> | |
| 5.6 Strategies for Recruitment and Retention | |
| 6. STUDY PRODUCT | |
| 6.1 Study Product(s) and Administration –Remdesivir, Risankizumab, and Placebo. | |
| 6.1.1 Study Product Description | |
| 6.1.2 Dosing and Administration | 18 |
| 6.1.3 Dose Escalation | |
| 6.1.4 Dose Modifications | |
| | 1 |

| Table 1. BET-A Schedule of Assessments | 6 |
|---|---|
| Table 2. Summary of Adverse Reaction Rates in Subjects with Mild, Moderate, or Severe | |
| COVID-19 in ACTT-1 | 9 |
| Table 3. BET-A Study Objectives | 10 |

#### 1. PROTOCOL SUMMARY

## 1.1 Synopsis

#### **Rationale for Proposed Clinical Study**

Studies have shown that moderate to severe cases of COVID-19 are characterized by marked inflammation and cytokine storm.(1-5) Over the course of the SARS-CoV2 pandemic, the T<sub>H</sub>17 pathway has specifically been identified as a potentially important contributor to disease pathophysiology.(6, 7) Evaluation of a patient with severe COVID-19 showed an increased concentration of T<sub>H</sub>17 cells in peripheral blood.(8) The role of T<sub>H</sub>17 immune responses in COVID-19 pathogenesis appears to be comparable to its roles in SARS and MERS.(9, 10)

In light of these data, drugs that inhibit T<sub>H</sub>17 immune responses hold promise for COVID-19 treatment. Since IL-23 has an essential role in the differentiation and expansion of T<sub>H</sub>17 cells, inhibition of IL-23 is expected to dampen COVID-19 immunopathogenesis.(11, 12) According to findings from The Inflammatory Bowel Diseases Surveillance Epidemiology of Coronavirus Under Research Exclusion (Secure-IBD) database,(13) patients on IL-12/-23 inhibitors had milder COVID-19 disease courses than those on most other classes of medication, with 116/139 (83%) managed as outpatients and only 5/139 (4%) meeting the combined endpoint of either ICU admission, mechanical ventilation or death (compared to 284/481 (59%) and 60/481 (12%) who were taking sulfasalazine or mesalamine for their baseline IBD control. This suggests that inhibition of the IL-23 pathway, at least early in infection, may be useful in modulating disease severity. Thus, we hypothesize that treatment of COVID-19 patients with risankizumab, an IL-23 antagonist, will improve clinical outcomes.

#### **Study Design**

See the Master protocol document for a description of the study design.

#### **Study Objectives**

See Table 3 in Section 3.

#### **Study Population**

This trial will study risankizumab in a hospitalized adult population (≥18 years old) with COVID-19. See Sections 5.1 and 5.2 for inclusion and exclusion criteria.

#### **Study Phase**

• Phase 2

#### **Study Sites**

There will be up to 70 domestic sites and 5 international sites.

#### **Study Interventions**

All subjects will receive remdesivir as a 200-mg intravenous (IV) loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose during hospitalization up to a maximum of 10 total doses (i.e., loading + maintenance doses received during study and pre-study if

Version 6 21 September 2021

Appendix A – BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir

applicable). The duration of dosing may be adjusted by the site similar to what is described in the product label and based on a subject's clinical course and ultimate disease severity.

In addition to receiving remdesivir, subjects in the BET-A stage will be randomized to receive risankizumab or placebo as follows:

- Risankizumab 1200-mg IV infusion once on Day 1.
- Placebo will be given at an equal volume at the same schedule.

#### **Study Duration**

This stage is anticipated to enroll over 3 months, with an additional 1 month of follow-up, and 2 months to lock the database.

#### **Participant Duration**

An individual subject will complete the study in about 60 days, from screening at Day -1 or 1 to completion of follow-up on Day  $60 \pm 3$  days.

#### **DSMB**

See Section 10.1.6.2 of the Master protocol document.

## 1.2 Schedule of Assessments

## Table 1. BET-A Schedule of Assessments

| | Screen | Baseline | Study Intervention Period | Follow-up Visits | | | | |
|---|---|---|---|---|---|---|---|---|
| Doy +/ Window | _1 on 1 | 115 | Daily until hospital | 810 | 15 <sup>6</sup> | <b>22</b> <sup>10</sup> | <b>29</b> <sup>6</sup> | $60^{10}$ |
| Day +/- window | Day +/- Window —1 or 1 | | discharge (up to Day 29) | ± 2 | ± 2 | ± 3 | ± 3 | ± 3 |
| ELIGIBILITY | | | | | | | | |
| Informed consent | X | | | | | | | |
| Demographics & Medical History | X | | | | | | | |
| Targeted physical exam | X | | | | | | | |
| Review SARS-CoV-2 results | X | | | | | | | |
| STUDY INTERVENTION | | | | | | | | |
| Randomization | | X | | | | | | |
| Administration of investigational agent | | <ul> <li>Risankizumab or placebo: one infusion on Day 1</li> <li>Remdesivir: IV daily for 5-10 days or until discharge.</li> </ul> | | | | | | |
| STUDY PROCEDURES | | | | | | | | |
| Vital signs and NEWS score 1, 14 | | $X^3$ | | | | | | |
| Clinical data collection <sup>1</sup> | | $X^3$ | Daily until discharge | X | X | X | X | $X^{13}$ |
| Adverse event evaluation | | $X^3$ | Daily until discharge | X | X | X | X | X |
| Concomitant medication review <sup>12</sup> | | $X^3$ | Day -7 until discharge | X | X | X | X | |
| | | - 11 | Buy / until disonalge | 11 | - 11 | | | |
| SAFETY LABORATORY | | | | | | | | |
| Safety hematology, chemistry, and liver tests <sup>4, 9</sup> | $X^2$ | $X^3$ | Day 3, 5, 8, 11 (all $\pm$ 1 day) if hospitalized <sup>5</sup> | | X | | X | |
| Pregnancy test for females of childbearing potential | X <sup>2</sup> | | | | | | | |
| RESEARCH LABORATORY <sup>16</sup> | | | | | | | | |
| Oropharyngeal swab <sup>7</sup> | | $X^3$ | Day 3, 5, 8, 11 (all $\pm$ 1 day) if hospitalized | | X | | X | |
| Blood draw for serum and plasma. Specific testing is as follows: | | $X^3$ | Day 3, 5, 8, 11 (all $\pm$ 1 day) if hospitalized | | X | | X | |
| PCR SARS-CoV-2 | | $X^3$ | Day 3, 5, 8, 11 (all $\pm$ 1 day) if hospitalized | | | | | |
| Proteomic analysis (including specifically for risankizumab IL-17A, IL-22, and IL-1b) | | $X^3$ | Day 3, 8, (all $\pm$ 1 day) if hospitalized | | X | | X | |
| Risankizumab<br>pharmacokinetics <sup>11</sup> | | $X^8$ | Day 5 (± 1 day) if<br>hospitalized | | X | | X | |
| Risankizumab<br>immunogenicity <sup>11</sup> | | X <sup>8</sup> | | | | | X | |
| Serum for secondary research | | $X^3$ | Day 3, 5, 8, 11 (all $\pm$ 1 day) if hospitalized. | | X | | X | |
| Blood for RNA | | $X^3$ | Day 3, 8 (all ± 1 day) if hospitalized | | X | | X | |
| Blood for PBMC <sup>11</sup> | | $X^3$ | Day 3, 8 (all ± 1 day) if hospitalized | | X | | X | |
| Notes: | | | | | | | | |

<sup>1</sup> Refer to Section 8.1 of the protocol for details of clinical data to be collected including ordinal score, NEWS, oxygen requirement, mechanical ventilator requirement, etc.

- <sup>2</sup> Screening laboratory tests include: ALT, AST, creatinine (and calculate an estimated glomerular filtration rate (eGFR) the formula used is determined by the sites, but should be consistent throughout the study), and urine or serum pregnancy test for females of child-bearing potential. Laboratory tests performed as part of routine clinical care in the 48 hours prior to enrollment will be accepted for determination of eligibility.
- <sup>3</sup> Baseline assessments should be performed prior to first infusion. Laboratory tests performed as part of routine clinical care in the 24 hours prior to first dose will be accepted for the baseline safety laboratory tests. Baseline may be the same as the screening laboratory tests if obtained in the 24 hours prior to first dose.
- <sup>4</sup> Safety laboratory tests include WBC with differential, hemoglobin, platelets, creatinine, total bilirubin, ALT, AST, and INR.
- <sup>5</sup> Any laboratory tests performed as part of routine clinical care within the specified visit window can be used for safety laboratory testing. <sup>6</sup> In-person visits are preferred but recognizing quarantine and other factors may limit the subject's ability to return to the site for the visit. In this case, the visit may be performed by phone.
  - If still hospitalized at Day 15 and 29 or returns for an in-person visit: assess adverse events, collect clinical data, vital signs, safety laboratory tests, and research laboratory samples (OP swab and blood) as able.
  - If phone call only on Days 15 and 29 and all Day 22 and Day 60 visits: assess adverse events, clinical status (ordinal scale), readmission to a hospital, and mortality only.
- <sup>7</sup> Oropharyngeal swabs are preferred, but if these are not obtainable, saliva or nasopharyngeal or nasal swabs may be substituted.
- <sup>8</sup> *Pre-dose serum sample collections for PK and immunogenicity.*
- <sup>9</sup> To include markers of inflammation and coagulation: CRP, ferritin, fibrinogen, d-dimer.
- <sup>10</sup> Day 8, 22 and 60 visits performed by phone call or home visit if discharged from the site hospital: assess adverse events, clinical status (ordinal scale), readmission to a hospital, and mortality only.
- <sup>11</sup> Only collected at selected sites capable of processing.
- <sup>12</sup> Steroids and other concomitant therapies intended as specific treatment of COVID-19, as well as all biologics, will be assessed from 7 days prior to enrollment to Day 29. All other concomitant medications will be assessed from 7 days prior to enrollment to Day 15 or upon discharge, whichever comes first.
- <sup>13</sup> Ordinal score only.
- <sup>14</sup> Vital signs include temperature, systolic blood pressure, heart rate, respiratory rate, O2 saturation and level of consciousness. In addition, height and weight are obtained only at baseline (height can be self-reported). Vital signs collected as part of standard care may be used
- <sup>15</sup> Day 1 is defined as the calendar day of randomization.
- <sup>16</sup> Blood draws for research labs may be omitted on any given study day if inappropriate for a subject's clinical status per site investigator judgment.

## 2. INTRODUCTION

## 2.1 Study Rationale

See Section 1.1 of this Appendix.

## 2.2 Background

## 2.2.1 Purpose of Study

See Section 1.1 of this Appendix.

#### 2.2.2 Potential Therapeutic Agents

Remdesivir is a broad-spectrum nucleotide prodrug that inhibits RNA-dependent RNA polymerase. Remdesivir is licensed for the treatment of COVID-19 requiring hospitalization. In the ACTT-1 trial, remdesivir has been demonstrated to decrease the time to recovery from 15 to 10 days (recovery rate ratio 1.29 (1.12 to 1.49); P<0.001).(14) All subjects in the trial will be given remdesivir.

Risankizumab is a humanized immunoglobulin G1 (IgG1) monoclonal antibody that antagonizes IL-23. It is indicated for the treatment of moderate-to-severe plaque psoriasis, and is currently under investigation in patients with ulcerative colitis, Crohn's disease, and hidradenitis suppurativa.

#### 2.3 Risk/Benefit Assessment

#### 2.3.1 Known Overall Risks

Potential risks of participating in this stage are those associated with having blood drawn, the IV catheterization, possible reactions to remdesivir and risankizumab (as noted in Sections 2.3.2-2.3.3), and breach of confidentiality.

Drawing blood may cause transient discomfort and fainting. Fainting is usually transient and managed by having the subject lie down and elevate his/her legs. Bruising at the blood collection sites may occur but can be prevented or lessened by applying pressure to the blood draw site for a few minutes after the blood is taken. IV catheterization may cause insertion site pain, phlebitis, hematoma formation, and infusate extravasation; less frequent but significant complications include bloodstream and local infections. The use of aseptic (sterile) technique will make infection at the site where blood will be drawn or at catheter site less likely. Rarely, severe allergic reactions (called anaphylaxis) can occur and may cause heart attacks and, if untreated, even death.

#### Risks to Privacy

Subjects will be asked to provide personal health information (PHI). All attempts will be made to keep this PHI confidential within the limits of the law. However, there is a chance that unauthorized persons will see the subject's PHI. All study records will be kept in a locked file cabinet or maintained in a locked room at the participating clinical site. Electronic files will be password protected. Only people who are involved in the conduct, oversight, monitoring, or auditing of this trial will be allowed access to the PHI that is collected. Any publication from this trial will not use information that will identify subjects. Organizations that may inspect and/or copy research records maintained at the participating site for quality assurance and data analysis include groups such as the IRB, NIAID and applicable regulatory agencies (e.g., FDA). For more information about confidentiality and privacy see Section 10.1.3 in the Master protocol document.

#### **Risks of Genetic Testing**

Genetic findings can have emotional and psychological consequences as well as implications for health, employability, and insurability for the subject and family members. However, state and federal laws provide protections against genetic discrimination. Samples and the resulting data will be coded and kept private. Additionally, to protect confidentiality, results will be entered into a password-protected database restricted to the PI or appointed designees. Genetic information would only be divulged if a subject signs a waiver on an insurance application. Study analyses will not result in discoveries about identity or paternity.

#### 2.3.2 Potential Risks of Remdesivir

Remdesivir is an FDA approved antiviral and may be obtained as part of standard care outside the clinical trial. For the purpose of the BET-A study, remdesivir is still considered a study product being used as part of an investigational trial and it will be tracked and monitored accordingly.

Transaminase elevations have been observed in healthy volunteers who received remdesivir; the transaminase elevations were mild (Grade 1) to moderate (Grade 2) in severity and resolved upon discontinuation of remdesivir. Transaminase elevations have also been reported in patients with COVID-19 who received remdesivir.

In ACTT-1, the collection of adverse event (AE) data in this trial was limited to severe (Grade 3) or potentially life-threatening (Grade 4) AEs, serious adverse events (SAEs), AEs leading to study drug discontinuation, and moderate (Grade 2) severity or higher hypersensitivity reactions. Rates of adverse reactions ( $\geq$  Grade 3), serious adverse reactions, and adverse reactions leading to treatment discontinuation are presented in Table 2.

Table 2. Summary of Adverse Reaction Rates in Subjects with Mild, Moderate, or Severe COVID-19 in ACTT-1

| Types of Adverse Reactions | Remdesivir N=532 n (%) | Placebo N=516 n (%) |
|------------------------------|------------------------|---------------------|
| Adverse reactions, Grades ≥3 | 41 (8%) | 46 (9%) |
| Serious adverse reactions | 2 (0.4%) <sup>a</sup> | 3 (0.6%) |
| Adverse reactions leading to | 11 (2%) <sup>b</sup> | 15 (3%) |
| treatment discontinuation | | |

a Seizure (n=1), infusion-related reaction (n=1).

There is the potential of the SARS-CoV-2 developing resistance to remdesivir, which could result in decreased efficacy. The clinical impact of the development of resistance is not clear at this time.

Coadministration of remdesivir and chloroquine phosphate or hydroxychloroquine sulfate is not recommended based on cell culture data demonstrating an antagonistic effect of chloroquine on the intracellular metabolic activation and antiviral activity of remdesivir.

See Package Insert for full discussion of clinical experience and risks.

#### 2.3.3 Potential Risks of Risankizumab

Potential risks include upper respiratory infection, fungal skin infection, headache, and tiredness. A total of 2234 subjects were treated with risankizumab in clinical studies for plaque psoriasis. In the first 16 weeks of treatment, infections occurred in 22.1% of the risankizumab group (90.8 events per 100 subject-years) compared to 14.7% of the placebo group (56.5 events per 100 subject-years) and did not lead to discontinuation of risankizumab. The rates of serious infections for both the risankizumab and placebo groups were ≤0.4%. Serious infections in the risankizumab-treated group included cellulitis, osteomyelitis, sepsis, and herpes zoster. In

b. Seizure (n=1), infusion-related reaction (n=1), transaminases increased (n=3), ALT increased and AST increased (n=1), GFR decreased (n=2), acute kidney injury (n=3).

ULTIMMA-1 and ULTIMMA-2 trials, through Week 52, the rate of infections (73.9 events per 100 subject-years) was similar to the rate observed during the first 16 weeks of treatment. Through Week 52, no new adverse reactions were observed, and the rates of the adverse reactions were similar to those identified during the first 16 weeks of treatment. During this time period, serious infections that led to study discontinuation included pneumonia.

In the Phase 2 ulcerative colitis study, 49% of patients treated with up to three doses of 1200 mg of risankizumab IV over a 3-month period and 41% of patients in the placebo arm were on concomitant steroids. There was no difference in the overall safety profile of patients that were on corticosteroid medication and received either risankizumab 1200 mg or placebo, indicating no safety concerns with concomitant use of risankizumab with steroids.

#### 2.3.4 Known Potential Benefits

Individual subjects with COVID-19 participating in this stage may or may not experience improved clinical outcomes. However, there is potential benefit to society from their participation in this study resulting from insights gained about the therapeutic agent under study as well as the natural history of the disease. While there may not be benefits for an individual subject, there may be benefits to society if a safe, efficacious therapeutic agent can be identified during this global COVID-19 outbreak.

#### 3. OBJECTIVES AND ENDPOINTS

**Table 3. BET-A Study Objectives** 

| OBJECTIVES | ENDPOINTS (OVERCOME AND A SUPPLIE) |
|---|---|
| | (OUTCOME MEASURES) |
| Primary | |
| To evaluate the clinical efficacy of risankizumab relative to the control arm in adults hospitalized with COVID-19 according to clinical status (8-point ordinal scale) at Day 8. | 1. Not hospitalized, no new or increased** limitations on activities; 2. Not hospitalized, but new or increased limitation on activities and/or requiring new or increased home oxygen, CPAP or BiPAP; 3. Hospitalized, not requiring new or increased supplemental oxygen - no longer requires ongoing medical care; 4. Hospitalized, not requiring new or increased supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5. Hospitalized, requiring new or increased supplemental oxygen; 6. Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices; 7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane |

ACTIV-5/Big Effect Trial (BET) Appendix A – BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir

| OBJECTIVES | ENDPOINTS<br>(OUTCOME MEASURES) |
|---|---|
| | oxygenation (ECMO);<br>8. Death. |
| Key Secondary | |
| 1. To evaluate the clinical efficacy of risankizumab as assessed by time to recovery compared to the control arm. | Day of recovery is defined as the first day on which the subject satisfies 1 of the following 3 categories from the ordinal scale (and does not return to a score of 4 or higher for the remainder of the study period): 1. Not hospitalized, no new or increased limitations on activities; 2. Not hospitalized, but new or increased limitation on activities and/or requiring new or increased home oxygen, CPAP, or BiPAP; 3. Hospitalized, not requiring new or increased supplemental oxygen - no longer requires ongoing medical care. |
| 2. To evaluate the proportion of subjects alive and without respiratory failure through Day 29. | Subjects in ordinal scale 5 or 6 at baseline who did not meet either of the following two categories at any point through Day 29: 7. Hospitalized, on invasive mechanical ventilation or ECMO; 8. Death. |
| Other Secondary | |
| <ol> <li>To evaluate the clinical efficacy of risankizumab as compared to the control arm as assessed by: <ul> <li>Clinical Severity</li> <li>Ordinal scale: <ul> <li>Clinical status using ordinal scale at Days 15 and 29.</li> <li>Time to an improvement of one category and two categories from Day 1 (baseline) using an ordinal scale.</li> <li>Mean change in the ordinal scale from Day 1 to Days 3, 5, 8, 11, 15, 22, and 29.</li> </ul> </li> </ul> </li> </ol> | Clinical outcome assessed using ordinal scale daily while hospitalized and on Days 15, 22, and 29. |
| <ul><li>Oxygenation:</li><li>Supplemental oxygen use up to Day</li></ul> | Days of supplemental oxygen (if applicable) up to Day 29. |

ACTIV-5/Big Effect Trial (BET) Appendix A – BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir

| OBJECTIVES | ENDPOINTS<br>(OUTCOME MEASURES) |
|---|---|
| 29. | |
| <ul> <li>Non-invasive ventilation/high-flow oxygen:</li> <li>Non-invasive ventilation/high-flow oxygen use up to Day 29.</li> <li>Incidence and duration of new non-invasive ventilation or high-flow oxygen use through Day 29.</li> </ul> | Days of non-invasive ventilation/high-<br>flow oxygen (if applicable) up to Day 29. |
| <ul> <li>Invasive Mechanical Ventilation/<br/>ECMO:</li> <li>Ventilator/ECMO use up to Day 29.</li> <li>Incidence and duration of new<br/>mechanical ventilation or ECMO<br/>use through Day 29.</li> </ul> | Days of invasive mechanical<br>ventilation/ECMO (if applicable) up to<br>Day 29. |
| <ul> <li>Proportion of subjects alive and<br/>without respiratory failure at Day 29.</li> </ul> | Proportion of subjects who did not meet either of the following two categories on Day 29: 7. Hospitalized, on invasive mechanical ventilation or ECMO; 8. Death. |
| <ul><li>Hospitalization:</li><li>Duration of hospitalization (days).</li></ul> | Days of hospitalization up to Day 29. |
| <ul> <li>Mortality:</li> <li>14-day mortality.</li> <li>29-day mortality.</li> <li>Time to death up to Day 29.</li> <li>60-day mortality.</li> </ul> | Date and cause of death (if applicable). |
| Markers of inflammation and coagulation. | C-reactive protein (CRP), ferritin, D-dimer, and fibrinogen on Day 1; Days 3, 5, 8, and 11 (while hospitalized); and Days 15 and 29 (if attends in-person visit or still hospitalized). |
| <ul> <li>2. To evaluate the safety of risankizumab as compared to the control arm as assessed by:</li> <li>Cumulative incidence of SAEs through Day 60.</li> <li>Cumulative incidence of Grade 3 and 4 clinical and/or laboratory AEs through Day 60.</li> </ul> | <ul><li>SAEs.</li><li>Grade 3 and 4 AEs.</li></ul> |

ACTIV-5/Big Effect Trial (BET) Appendix A – BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir

| OBJECTIVES | ENDPOINTS<br>(OUTCOME MEASURES) |
|---|---|
| <ul> <li>Discontinuation or temporary suspension of study product administration (for any reason).</li> <li>Changes in white blood cell (WBC) count with differential, hemoglobin, platelets, creatinine, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and international normalized ratio (INR) over time (analysis of lab values in addition to AEs noted above).</li> </ul> | <ul> <li>Episodes of early discontinuation or interruption of study product administration.</li> <li>WBC with differential, hemoglobin, platelets, creatinine, total bilirubin, ALT, AST, and INR on Day 1; Days 3, 5, 8, and 11 (while hospitalized); and Days 15 and 29 (if attends in-person visit or still hospitalized).</li> </ul> |
| Exploratory | |
| <ol> <li>To evaluate the virologic efficacy of risankizumab as compared to the control arm as assessed by: <ul> <li>Percent of subjects with SARS-CoV-2 detectable in saliva (or best technology) sample at Days 3, 5, 8, 11, 15, and 29.</li> <li>Quantitative SARS-CoV-2 virus in saliva (or best technology) sample at Days 3, 5, 8, 11, 15, and 29.</li> <li>Quantitative SARS-CoV-2 virus in blood at Days 3, 5, 8, and 11.</li> </ul> </li> </ol> | <ul> <li>Qualitative and quantitative polymerase chain reaction (PCR) for SARS-CoV-2 in OP swab on Day 1; Days 3, 5, 8, and 11 (while hospitalized); and Days 15 and 29 (if attends in-person visit or still hospitalized).</li> <li>Qualitative and quantitative PCR for SARS-CoV-2 in blood on Day 1; Days 3, 5, 8, and 11 (while hospitalized).</li> </ul> |
| 2. To evaluate the impact of study interventions on markers of inflammation and immune response. | <ul> <li>Proteomic analysis of plasma cytokines and markers of inflammation including IL-17A, IL-22 and IL-1b.</li> <li>Transcription, epigenetic, and molecular profiles of mRNA in peripheral blood mononuclear cells (PBMC).</li> <li>Phenotypic and responsiveness markers in PBMC.</li> </ul> |
| 3. To evaluate post-baseline usage of key concomitant COVID-19 treatments (e.g., steroids) in investigational therapeutic arms as compared to the control arm. | Use of concomitant COVID-19 treatments up to Day 29. |

| OBJECTIVES | | ENDPOINTS<br>(OUTCOME MEASURES) | |
|---|---|---|---|
| Stage-specific<br>objective/endpoint | 4. To evaluate risankizumab pharmacokinetics (PK) and immunogenicity in subjects with COVID-19. | • | Serum samples for PK (at pre-dose, Day 5, Day 15, and Day 29) and serum samples for anti-drug antibodies and neutralizing antibodies at pre-dose and Day 29. |

<sup>\*\* &</sup>quot;New or increased" is relative to pre-COVID status

#### 4. STUDY DESIGN

## 4.1 Overall Design

See Section 1.1 of the Master protocol document.

#### **4.2 Justification for Dose**

#### **4.2.1 Justification for Dose of Remdesivir**

The dose of remdesivir used in this study will be the same dose shown to be efficacious in the ACTT-1 clinical trial,(14) and are the US FDA approved doses. The duration of dosing may be adjusted by the site according to clinical severity. The maximum number of doses to be given during hospitalization is ten doses. This includes the loading dose and all maintenance doses given during the study and pre-study if applicable.

#### 4.2.2 Justification for Dose of Risankizumab

The dose of risankizumab used in this stage will be 1200 mg administered as a single dose intravenously (IV). This is the same dose level as the highest dose used in the multiple dose induction Phase 3 clinical trials for inflammatory bowel diseases. The 1200 mg IV dose given once every 4 weeks for 3 doses has been evaluated in a dose-ranging Phase 2 clinical study in subjects with UC

Phase 3 study in subjects with CD. Available data from these studies showed that the 1200 mg risankizumab dose is well tolerated and dose-ranging data including higher and lower doses did not reveal any exposure-dependent safety issues. Therefore, given the novel setting of COVID-19 and the acute nature of the disease onset in the target patient population of the study, 1200 mg IV is selected to provide best opportunity for efficacy in this POC study. The dose is expected to be safe and well tolerated in COVID-19 patients. It is also expected to provide a quick onset of drug exposure following IV administration and duration of exposure long enough to cover the 29 days of the main study thanks to the long elimination half-life (approximately 28 days) of risankizumab.

## 5. STUDY POPULATION

Approximately 200 (100 treatment and 100 shared placebo) male and non-pregnant female adults ≥18 years of age or older with COVID-19 and who meet all eligibility criteria will be enrolled at up to 70 domestic sites and 5 international sites. The target population should reflect the community at large. The estimated time from screening (Day -1 or Day 1) to end of study for an individual subject is approximately 60 days.

Subject inclusion and exclusion criteria must be confirmed by a clinician named on the delegation log. If there is any uncertainty, the site PI may consult the DMID Medical Officer on whether a potential subject is eligible for study enrollment; the site PI is ultimately responsible for making the final decision. There is no exclusion for receipt of SARS-CoV-2 vaccine (experimental or licensed).

#### 5.1 Inclusion Criteria

- 1. Admitted to a hospital with symptoms suggestive of COVID-19 and requires ongoing medical care.
- 2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
- 3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
- 4. Male or non-pregnant female adult  $\geq$ 18 years of age at time of enrollment.
- 5. Illness of any duration and has laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other commercial or public health assay (e.g., Nucleic Acid Amplification Test [NAAT], antigen test) in any respiratory specimen or saliva ≤14 days prior to randomization.
- 6. Illness of any duration, and requiring, just prior to randomization, supplemental oxygen (any flow), mechanical ventilation or ECMO (ordinal score 5, 6, or 7).
- 7. Women of childbearing potential must agree to either abstinence or use at least one acceptable method of contraception from the time of screening through 5 months post study IP dosing.

Note: Acceptable methods include barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUDs), hormonal contraceptives, oral contraceptive pills, and surgical sterilization.

8. Agrees not to participate in another blinded clinical trial (both pharmacologic and other types of interventions) for the treatment of COVID-19 through Day 29 (see Section 5.4 for more information about concurrent trial participation).

#### 5.2 Exclusion Criteria

- 1. ALT or AST > 5 times the upper limit of normal.
- 2. Subjects with a low glomerular filtration rate (eGFR), specifically:
  - a. Subjects with an eGFR 20-30 mL/min are excluded unless in the opinion of the PI, the potential benefit of participation outweighs the potential risk of study participation.
  - b. All subjects with an eGFR <20 mL/min (including hemodialysis and hemofiltration) are excluded.

- 3. Pregnancy or breast feeding.
- 4. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours of enrollment.
- 5. Allergy to any study medication.
- 6. Received five or more doses of remdesivir prior to screening.
- 7. Received two or more doses of > 60 mg of prednisone or equivalent in the 7 days prior to screening
- 8. Received small molecule tyrosine kinase inhibitors, including Janus kinase (JAK) inhibitors (e.g., baricitinib, ibrutinib, acalabrutinib, imatinib, gefitinib), in the 4 weeks prior to screening.\*
- 9. Received monoclonal antibodies targeting cytokines (e.g., TNF inhibitors, anti-IL-1 [e.g., anakinra, canakinumab], anti-IL-6 [e.g., tocilizumab, sarilumab, sitlukimab]), or T-cells (e.g., abatacept) in the 4 weeks prior to screening.\*
- 10. Received monoclonal antibodies targeting B-cells (e.g., rituximab, and including any targeting multiple cell lines including B-cells) in the 3 months prior to screening.\*
- 11. Received GM-CSF agents (e.g., sargramostim) within 2 months prior to screening.\*
- 12. Received other immunosuppressants in the 4 weeks prior to screening and in the judgment of the investigator, the risk of immunosuppression with risankizumab is larger than the risk of COVID-19.\*
- 13. Received any live vaccine in the 4 weeks prior to screening.
- 14. Known active tuberculosis.
- 15. Known history of HIV, Hepatitis B (HBV) or untreated hepatitis C (HCV) infection.
- 16. History of pulmonary alveolar proteinosis (PAP).\*
- 17. Has a malignancy and currently receiving immunosuppressive chemotherapy, immunodeficiency, uncontrolled opportunistic infection, or uncontrolled cirrhosis.
- 18. Has a medical condition that could, in the judgment of the investigator, limit the interpretation and generalizability of trial results.
- 19. Positive test for influenza virus during the current illness (*influenza testing is not required by protocol*).
- 20. Previous participation in an ACTIV-5/BET trial.

#### \* Stage-specific criteria.

#### **5.2.1** Exclusion of Specific Populations

Children and adolescents will not be included in this trial. Remdesivir has only been used in a small number of pediatric patients. Initial information about the epidemiology of COVID-19 indicates that the overwhelming burden of severe disease occurs among older adults, especially those with comorbidities. The safety and efficacy of risankizumab in pediatric patients less than 18 years of age have not yet been established. Given significant gaps in knowledge in this population, and a low incidence of severe morbidity/mortality in children, the risk/benefits do not warrant inclusion of this population into this trial at this time.

Remdesivir and risankizumab have not been studied in pregnant women. Because the effects on the fetus and the pregnant woman are not fully known, pregnant women will not be eligible for the trial.

It is not known whether remdesivir or risankizumab is secreted in human milk. Because the effects of remdesivir and risankizumab on the breastfeeding infant is not known, women who are breast feeding will not be eligible for the trial.

## 5.3 Inclusion of Vulnerable Subjects

Certain human subjects are categorized as vulnerable populations and require special treatment with respect to safeguards of their well-being. For this clinical trial, examples include cognitively impaired or mentally disabled persons and intubated individuals who are sedated. When it is determined that a potential research subject is cognitively impaired, federal and institutional regulations permit researchers to obtain consent from a legally authorized representative (LAR). The study team will obtain consent from these vulnerable subjects using an IRB-approved protocol-specific process for consent using a LAR.

For subjects for whom a LAR gave consent, during the course of the study, if the subject regains the capacity to consent, informed consent must be obtained from the subject and the subject offered the ability to leave the study if desired.

## 5.4 Lifestyle Considerations

During this study, subjects are asked to:

- Refrain from drinking alcohol through Day 15.
- Avoid getting pregnant during the study from the time of screening through 5 months post study IP dosing.
- Subject's participation in other trials for COVID-19 or SARS-CoV-2 infection are restricted/permitted as follows:
  - Blinded trials of interventions of antiviral or immunomodulatory agents for treatment of COVID-19 are prohibited through Day 29.
  - Co-enrollment in non-blinded (open-label) interventional studies that evaluate how to apply a standard of care intervention or strategy for patients with COVID-19 (e.g., comparing dose, duration or schedule of VTE prophylaxis regimens; ICU strategies such as proning, etc.) is permitted.
  - Co-enrollment in natural history studies of COVID-19 and/or studies of SARS-CoV-2 diagnostics is permitted.
  - o Participation in both ACTIV-5/BET and these studies can only occur if the recommended blood collection volumes are not exceeded.
  - If a subject is co-enrolled in a prohibited study noted above, this should be reported as a protocol deviation, but the subject should not be withdrawn from this trial to participate in the other study. Full follow-up should occur per protocol.

#### 5.5 Screen Failures

Following consent, after the screening evaluations have been completed, the investigator or designee is to review the inclusion/exclusion criteria and determine the subject's eligibility for the study stage. If there is any uncertainty, the PI should make the decision on whether a potential subject is eligible for study enrollment.

Only basic demographic information and the reason(s) for ineligibility will be collected on screen failures. Subjects who are found to be ineligible will be told the reason(s) for ineligibility.

Individuals who do not meet the criteria for participation in this study (screen failure) because of an abnormal laboratory finding may be rescreened once.

#### 5.6 Strategies for Recruitment and Retention

See Section 5.4 of the Master protocol document.

#### 6. STUDY PRODUCT

## 6.1 Study Product(s) and Administration –Remdesivir, Risankizumab, and Placebo

#### **6.1.1 Study Product Description**

#### Remdesivir Component:

Remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the solution and lyophilized formulations of remdesivir contains the following inactive ingredients: water for injection (solution only), betadex sulfobutyl ether sodium, and hydrochloric acid and/or sodium hydroxide.

#### Risankizumab Component:

Risankizumab is a humanized immunoglobulin (Ig) G1 antagonistic monoclonal antibody (mAb) directed against the p19 subunit of the human cytokine interleukin-23. Risankizumab is formulated in a buffer of 4.4 mM disodium succinate hexahydrate/succinic acid, 225 mM sorbitol, 0.2 mg/mL polysorbate 20, and WFI in a 6R vial.

Risankizumab matching placebo solution for infusion is available in a 6R vial containing Disodium Succinate, Succinic Acid, Sorbitol, Polysorbate 20, and water for injection with a pH of 6.2

#### 6.1.2 Dosing and Administration

All subjects will receive remdesivir as a 200 mg IV loading dose on Day 1, followed by a 100 mg once-daily IV maintenance dose for the duration of the hospitalization up to a 10-day total course. If subjects already received the loading dose prior to study enrollment, then start at 100 mg/day on Day 1. Any doses of remdesivir given within 1 week of enrollment will be counted, so that the total duration of remdesivir (i.e. pre-enrollment + on this trial) is up to 10 days (i.e., a maximum of 10 total infusions). Any doses of remdesivir were administered prior to study

enrollment should be documented in on the eCRF as a concomitant medication given prior to Day 1. The duration of dosing may be adjusted by the site similar to what is described in the package insert and based on a subject's clinical course and ultimate disease severity.

Any dose of remdesivir that is delayed may be given later that calendar day. Any dose or remdesivir that is missed (not given that calendar day) is not made up. The treatment course continues as described above even if the subject becomes PCR negative.

In addition to receiving remdesivir, subjects in the BET-A trial will be randomized to receive risankizumab or placebo as follows:

- Risankizumab 1200-mg IV infusion (300 mg x 4 vials) once on Day 1.
- Placebo will be given at an equal volume at the same schedule.

At least 20 minutes between administration of remdesivir and risankizumab or placebo are preferred if possible (to allow attribution of any infusion related adverse reactions). However, timely administration of both products is most important, and if the interval between products is likely to cause delays for either products, it can be omitted. See MOP for details.

If the dose of risankizumab is delayed, it should be given as soon as practical.

#### 6.1.3 Dose Escalation

Not Applicable

#### **6.1.4 Dose Modifications**

#### Remdesivir component:

The infusion should be held and not given if the subject is found to have any of the following laboratory values:

- eGFR decreases to < 20 mL/min
  - o Remdesivir infusion will resume when the eGFR increases to  $\geq 20$  mL/min and the potential benefit of giving remdesivir outweighs the potential risk.
  - o If renal function worsens during the study to the point that they require hemodialysis or hemofiltration, remdesivir will be discontinued.
- ALT and/or AST increases to > 5 times upper limits of normal (ULN); resume remdesivir infusions when ALT and AST ≤ 5 times ULN.

Risankizumab component: No dosing adjustment needed.

#### 6.1.5 Overdosage

There is no known antidote for remdesivir. In the case of overdose, the subject should receive supportive therapy based on the subject's signs and symptoms.

In the event of risankizumab overdosage, monitor the patient for any signs or symptoms of adverse reactions and administer appropriate symptomatic treatment immediately.

## 6.2 Preparation/Handling/Storage/Accountability

#### 6.2.1 Acquisition and Accountability

Investigational products (IP) will be shipped to the site either directly from participating companies, from the Sponsor, or from other regional or local drug repositories. All other supplies should be provided by the site. Multiple lots of each IP may be supplied.

Study products received at the sites will be open label and not kit specific, unless specified in the stage-specific Manual of Procedures (MOP). Drug preparation will be performed by the participating site's research pharmacist on the same day of administration to the subject. See the MOP for detailed information on the preparation, labeling, storage, and administration of remdesivir, risankizumab, and placebo.

#### **Accountability**

The site PI is responsible for study product distribution and disposition and has ultimate responsibility for study product accountability. The site PI may delegate to the participating site's research pharmacist responsibility for study product accountability. The participating site's research pharmacist will be responsible for maintaining complete records and documentation of study product receipt, accountability, dispensation, storage conditions, and final disposition of the study product(s). Time of study drug administration to the subject will be recorded on the appropriate data collection form (CRF). All study product(s), whether administered or not, must be documented on the appropriate study product accountability record or dispensing log. The Sponsor's monitoring staff will verify the participating site's study product accountability records and dispensing logs per the site monitoring plan. Refer to the protocol-specific MOP for details on storing study medications.

#### **Destruction**

After the study treatment period has ended or as appropriate over the course of the study after study product accountability has been performed, used active and placebo vials can be destroyed on-site following applicable site procedures with a second staff member observing and verifying the destruction.

Unused vials at the end of the study should be saved until instructed by the Sponsor.

#### 6.2.2 Formulation, Appearance, Packaging, and Labeling

#### **Remdesivir component**

Remdesivir may be supplied in two formulations:

• The concentrated solution of remdesivir is supplied as a single dose in a Type 1 clear glass vial containing 100 mg/20 mL (5 mg/mL) of remdesivir per vial for dilution into 0.9% sodium chloride infusion bag. It is a sterile, preservative-free, clear, colorless to yellow, aqueous-based concentrated solution that is to be diluted into 0.9% sodium chloride infusion bag prior to administration by intravenous infusion. In addition to the active ingredient, the solution formulation of remdesivir contains the following inactive ingredients: water for injection, betadex sulfobutyl ether sodium, hydrochloric acid, and/or sodium hydroxide. For more information, refer to the MOP.

• The lyophilized formulation of remdesivir is a sterile, preservative-free, white to off-white to yellow powder containing 100 mg of remdesivir to be reconstituted with 19 mL of sterile water for injection and diluted into IV infusion fluids prior to IV infusion. Following reconstitution, each vial contains a 5 mg/mL remdesivir concentrated solution with sufficient volume to allow withdrawal of 20 mL (100 mg of remdesivir). It is supplied in a single-use, Type 1 clear glass vial. In addition to the active ingredient, the lyophilized formulation of remdesivir contains the following inactive ingredients: water for injection, betadex sulfobutyl ether sodium, hydrochloric acid, and/or sodium hydroxide. For more information, refer to the MOP.

Remdesivir will be labeled according to manufacturer specifications.

Risankizumab component

Risankizumab is a sterile isotonic aqueous solution for IV administration contained . Risankizumab drug product is a colorless to slightly yellow, clear to slightly opalescent solution, with an

#### **Placebo**

The supplied matching placebo of risankizumab is identical in physical appearance to the active IV formulation and contains the same inactive ingredients. The IV formulation of matching placebo is filled in a

. Each single-use vial

contains sufficient volume to allow withdrawal of 3.3 mL of placebo.

Each of the study products will be labeled according to manufacturer specifications and include the statement "Caution: New Drug Limited by Federal Law to Investigational Use."

#### 6.2.3 Product Storage and Stability

Refer to the MOP for instructions regarding the stability and storage of remdesivir, risankizumab, and placebo.

#### 6.2.4 Preparation

Refer to the MOP for details about preparation and handling of remdesivir, risankizumab, and placebo.

Remdesivir and risankizumab do <u>not</u> meet the criteria for a hazardous compound as defined by NIOSH and ASHP hazard classification systems. The study products may be prepared in a clean room but do not need to be prepared or handled in a fume hood.

Measures that minimize drug contact with the body should always be considered during handling, preparation, and disposal procedures as indicated in the MOP.

## 6.3 Measures to Minimize Bias: Randomization and Blinding

Randomization will be a two-step process. Patients will first be randomized to one of the stages to which they are eligible (e.g., risankizumab or other interventions) with equal allocation. Then

Protocol 20-0013A Version 6 ACTIV-5/Big Effect Trial (BET) 21 September 2021

Appendix A – BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir

patients are randomized to the active or placebo version of that intervention with allocation k:1, where k is the number of eligible stages the study site is currently randomizing. All eligible subjects will receive backbone therapy comprising remdesivir. Patients randomized to risankizumab in the first stage will be randomized to receive either risankizumab/remdesivir or placebo/remdesivir in the second stage. Randomization will be stratified by:

- Site
- Severity of illness at enrollment: baseline Ordinal Score 5 versus Ordinal Score 6 or 7 combined

The randomization procedure will be described in the MOP.

## **6.4** Study Intervention Compliance

Each dose of study product will be administered by a blinded member of the clinical research team who is qualified and licensed to administer the study product. Administration and date, and time, will be entered into the case report form (CRF).

## 6.5 Concomitant Therapy

#### 6.5.1 Permitted Concomitant Therapy and Procedures

For patients that are eligible for the study, other therapy received prior to enrollment with any other experimental treatment or off-label use of marketed medications that are intended as specific treatment for COVID-19 or the SARS-CoV-2 infection (i.e., post-exposure prophylaxis [PEP]) are permitted but must be discontinued on enrollment. There is no waiting period between discontinuation of these treatments and administration of study products. However, these prior treatments and their end date should be documented on the concomitant medication form in the EDC system.

Steroids for the treatment of COVID-19 may be used per the local institution's written standard of care (i.e., not just an individual clinician decision) or NIH COVID-19 Treatment Guidelines (https://www.covid19treatmentguidelines.nih.gov/). NIH COVID-19 Treatment Guidelines provide current evidence-based information about the optimal management of COVID-19. NIH COVID-19 Treatment Guidelines were updated on June 25, 2020 to include a Grade AI recommendation for using dexamethasone (6 mg per day for up to 10 days) in patients with COVID-19 who are mechanically ventilated and a Grade B1 recommendation for patients with COVID-19 who require supplemental oxygen but who are not mechanically ventilated based on preliminary data from the RECOVERY trial. The NIH Guidelines also recommend against using dexamethasone in COVID-19 patients who do not require supplemental oxygen.

Steroid regimens for other standard indications including asthma exacerbation, ARDS, COPD, laryngeal edema, adrenal insufficiency, shock, etc. are allowable up to a maximum of prednisone 60 mg daily or equivalent. All steroid use regardless of indication until Day 29 will be recorded in the EDC system.

Subjects who are taking another antiviral for a concurrent infection (e.g. oseltamivir for an influenza virus) or another existing medical condition (e.g. hydroxychloroquine for lupus) may

21 September 2021

Version 6

continue with the treatment. Note that these treatments may be thought of as an off-label medication for COVID-19, however, because they were being used prior to study enrollment for another indication, they are allowable.

Outpatient experimental treatment or off-label use of marketed medications that are intended as specific treatment for COVID-19 do not need to be discontinued if there is a written policy or guideline for the local standard of care and treatment of COVID-19 patients or SARS-CoV-2 infection (i.e., not just an individual clinician decision). In the absence of a local written standard of care, the National Institutes of Health (NIH) COVID-19 Treatment Guidelines may be used. If concomitant medications are used, there should be plans on how the concomitant drugs are stopped in case of additive toxicities.

Steroids and other concomitant therapies intended as specific treatment of COVID-19, as well as all biologics, will be assessed from 7 days prior to enrollment to Day 29. All other concomitant medications will be assessed from 7 days prior to enrollment to Day 15 or upon discharge, whichever comes first. All prescription medications should be recorded during this time period with the exceptions listed in the bullets below. All medications, except biologics, convalescent plasma and corticosteroids, can be recorded once regardless of the number of times it was given during the time period. For example, vasopressors should be recorded when first dose given (as the start date) and the last dose given (as the end date) during the period of assessment.

#### Sites do not need to record any of the following categories of medications as concomitant medications:

- o All topical medications: ointments, creams, and lotions;
- o All intranasal medications: nasal decongestants, nasal allergy medications, nasal steroids, and nasal saline drops/sprays;
- o All ophthalmic medications: ophthalmic allergy medication, ophthalmic medications for infection, and ophthalmic medications for eye dryness (e.g., saline eye drops);
- o Antiseptic mouth wash, lozenges;
- o Cough medication: mucolytics, cough suppressants, and expectorates;
- o GI medications: H2 blockers, proton pump inhibitors, GI stimulants, prokinetics, laxatives, stool softeners, antacids, anti-diarrheal and anti-nausea medications;
- o Insulin and medications for diabetic control;
- Symptomatic care medications: antipyretics, antihistamines, decongestants, and NSAIDs;
- O Vitamins, minerals or herbal supplements, dietary supplements, iron/ferrous sulfate, magnesium, calcium, electrolyte replacement;
- Albumin infusions:
- Melatonin;
- o Nicotine patch, lozenge, gum, or nasal spray, or other product to treat tobacco dependence;
- o Dyes: iodine-based dye, barium sulfate, and diatrizoate sodium.

See the MOP for more information about recording concomitant medications.

Protocol 20-0013A Version 6 ACTIV-5/Big Effect Trial (BET) 21 September 2021

Appendix A – BET-A: Risankizumab/Remdesivir vs. Placebo/Remdesivir

#### 6.5.2 Prohibited Concomitant Therapy

Receipt of any exclusionary treatments or medications prior to screening will be assessed at screening to determine eligibility as described in the exclusion criteria.

The following medications are prohibited during this study:

- Small molecule tyrosine kinase inhibitors (e.g., baricitinib, ibrutinib, acalabrutinib, imatinib, gefitinib).
- Monoclonal antibodies targeting cytokines (e.g., TNF inhibitors, anti-IL-1 [e.g., anakinra, canakinumab], anti-IL-6 [e.g., tocilizumab, sarilumab, sitlukimab]), or T-cells (e.g., abatacept).
- Monoclonal antibodies targeting B-cells (e.g., rituximab, and including any targeting multiple cell lines including B-cells).
- GM-CSF agents (e.g., sargramostim).
- Other immunosuppressants which, in the judgment of the investigator, pose risk of immunosuppression in combination with risankizumab that is larger than the risk of COVID-19.
- Chloroquine or hydroxychloroquine use for the treatment of COVID-19

A recent study found that chloroquine antagonizes remdesivir in a dose dependent manner as evidenced by an increase in the median effective dose (EC50) for remdesivir with increasing chloroquine concentration. Another in vitro study found that chloroquine induces a dose dependent inhibition of the formation of the active nucleoside triphosphate metabolite of remdesivir. Thus, chloroquine or hydroxychloroquine use for the treatment of COVID-19 is prohibited during the study.

Concomitant use of any other experimental treatment or off-label use of marketed medications intended as specific treatment for COVID-19 or SARS-CoV-2 infection, and not specified in local written guidelines or the NIH COVID-19 Treatment Guidelines are prohibited.

Overall, the risk of potential drug-drug interactions between risankizumab and concomitant medications is low. As a monoclonal antibody, risankizumab is not expected to undergo metabolism by hepatic enzymes or renal elimination. Drug interactions between risankizumab and substrates/inhibitors/inducers of drug metabolizing enzymes are not expected. Drugs with immunosuppressant effects such as methotrexate might reduce the immunogenicity to risankizumab but given the short duration of the study and the single dose administration, the potential impact of reduced immunogenicity on risankizumab safety or efficacy is expected to be low.

#### 6.5.3 Rescue Medicine

Not Applicable

#### 6.5.4 Non-Research Standard of Care

Not Applicable

#### 7. STUDY INTERVENTION DISCONTINUATION AND

## SUBJECT DISCONTINUATION/WITHDRAWAL

## 7.1 Halting Criteria and Discontinuation of Study Intervention

## 7.1.1 Individual Infusion Halting

See Section 6.1.4 for information about dosing modifications due to laboratory abnormalities.

For an individual subject, an individual infusion must be stopped if they have a suspected drug-related event of hypersensitivity (Grade 2 or higher) during the infusion. While there are no criteria for grading "hypersensitivity" in the Division of AIDS (DAIDS) Table for Grading the Severity of Adverse Events,(15) sites should use Acute Allergic Reaction from that toxicity table. Subjects who have an IV infusion stopped for a safety related issues will not continue with dosing.

The treatment of any given subject may be stopped for SAEs, clinically significant AEs, severe laboratory abnormalities, or any other medical conditions that indicate to the site Investigator that continued dosing is not in the best interest of the patient.

In addition, a subject in this clinical study may discontinue study drug at their request for any reason. Every effort should be made to encourage subjects to remain in the study for the duration of their planned outcome assessments. Subjects should be educated on the continued scientific importance of their data, even if they discontinue study drug.

Unless the subject withdraws consent, those who discontinue study drug early will remain in the study. The reason for subject discontinuation of study drug should be documented in the case report form.

#### 7.1.2 Study Halting

Given the potential severity of COVID-19, there are no pre-specified study stopping rules. Instead there will be close oversight by the protocol team and frequent DSMB reviews of the safety data.

## 7.2 Withdrawal from the Study

See Section 7.2 of the Master protocol document.

#### 7.3 Readmission

See Section 7.3 of the Master protocol document.

## 7.4 Lost to Follow-Up

See Section 7.4 of the Master protocol document.

## 8. STUDY ASSESSMENTS AND PROCEDURES

## 8.1 Screening and Efficacy Assessments

#### **8.1.1** Screening Procedures

Screening procedures may be done from Day -1 to Day 1 (Day 1 is the calendar day of randomization). However, in many cases all the screening assessments can be done in less than 24 hours. If that is the case, Day 1 pre-study product administration baseline assessments, specimen collection and the initial study product administration can occur on the same calendar day as the screening procedures.

After the informed consent, the following assessments are performed to determine eligibility:

- Confirm the positive SARS-CoV-2 test result (per inclusion criteria).
- Confirm that patient does not have a positive influenza test during the current illness for which they are being screened. (Influenza testing is not required per protocol.)
- Take a focused medical history, including the following information:
  - Day of onset of COVID-19 signs and symptoms.
  - Prior enrollment in ACTIV-5/BET.
  - History of vaccinations within 4 weeks prior to screening, including SARS-CoV-2 vaccination.
    - Exclusionary vaccine history includes any live vaccine (that is, live attenuated) within 4 weeks prior to screening.
  - History of chronic medical conditions, including chronic oxygen requirement and/or use of CPAP or BiPAP at home, prior to onset of COVID-19.
  - History of medication allergies.
  - Medications and therapies for this current COVID-19 illness and history of any medication listed in the exclusion criteria. Site should identify if the patient received any steroids in the 7 days prior to randomization.
  - Ask if the patient is participating in another clinical trial or plans to enroll in another clinical trial in the next 30 days.
- Women of childbearing potential must agree to either abstinence or use at least one
  acceptable method of contraception from the time of screening through 5 months post study
  IP dosing.\*
  - \*Note: Acceptable methods include barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUDs), hormonal contraceptives, oral contraceptive pills, and surgical sterilization.
- Targeted physical examination (targeted exam details in MOP).
- Height and weight (height can be self-reported).
- Assess need for supplemental oxygen, mechanical ventilation, or ECMO.
- Blood for screening laboratory evaluations, if not done as part of routine clinical care in the preceding 48 hours, should be collected to evaluate the following parameters:

- ALT
- AST
- Serum creatinine (and calculate eGFR)
  - Any automated calculation by the clinical laboratory or published formula for this calculation is acceptable. The site should select a formula to be used for all subjects enrolled at the site for the duration of the study.
- Urine or serum pregnancy test (in women of childbearing potential).

Clinical screening laboratory evaluations will be performed locally by the site laboratory. A screening lab (i.e., from the hematology and chemistry laboratory panels) may be repeated once if, in the opinion of the investigator, the laboratory abnormality is due to an intercurrent transient condition or it is an aberrant laboratory value. The overall eligibility of the subject to participate in the study will be assessed once all screening values are available. If performed just prior to randomization, data obtained from screening can also be a baseline assessment of severity and efficacy.

Study subjects who qualify will be randomized in the interactive response technology (IRT) system, and all others will be registered as screen failures only in the EDC system. The ordinal scale should be done at the time of randomization; the site will need this data to randomize the subject. The study team has 24 hours to complete other Day 1 baseline assessments prior to the first study product administration including the collection of the OP swab and blood, assessment of the ordinal scale and NEWS, and completing or recording a baseline physical examination that was done. Clinical laboratory tests performed as part of routine clinical care in the 48 hours prior to enrollment will be accepted for determination of eligibility.

#### 8.1.2 Efficacy Assessments

For all baseline assessments and follow-up visits, refer to the Schedule of Assessments (SOA) for procedures to be completed, and details below for each assessment.

Laboratory tests performed as part of routine clinical care in the 24 hours prior to first dose will be accepted for the baseline laboratory tests. Baseline may be the same as the screening laboratory tests if obtained in the 24 hours prior to first dose.

#### 8.1.2.1 Measures of Clinical Support, Limitations, and Infection Control

The subject's clinical status will be captured on each study day while hospitalized up until and including Day 29. Once subjects are discharged from the hospital, they will have a study visit on Days 8, 15, 22, 29, and 60 visits (only the ordinal score will be obtained on Day 60) as an outpatient. The Day 8, Day 22 and Day 60 visits do not have laboratory tests or collection of samples and may be conducted by phone. Day 15 and 29 visits are preferred to be in person in order to collect safety laboratory testing, stored samples, and virologic assessments but may be performed. Clinical status is largely measured by the ordinal scale. The ordinal scale can also be evaluated over the phone if the discharged subject is unable to return for in-person visits on Day 15 and 29.

The following measures are recorded for the ordinal scale. See MOP for more detailed description of ventilatory devices in each category:

- Hospitalization.
- Oxygen requirement.
- Non-invasive mechanical ventilation (via mask) requirement.
- High-flow oxygen requirement.
- Invasive mechanical ventilation (via endotracheal tube or tracheostomy tube) requirement.
- ECMO requirement.
- Ongoing medical care preventing hospital discharge (COVID-19 related or other medical conditions).
- Limitations of physical activity (self-assessed and reported as new or increased limitations as compared to status prior to the onset of COVID-19).
- Isolated for infection control purposes.

#### 8.1.2.2 Ordinal Scale

The ordinal scale is the primary measure of clinical outcome per the Master protocol document (Section 8.1.1.1).

#### **8.1.3** Exploratory Assessments

See Section 8.1.2 of the Master protocol document. Additional exploratory assessments include:

- Qualitative and quantitative polymerase chain reaction (PCR) for SARS-CoV-2 in OP swab on Day 1; Days 3, 5, 8, and 11 (while hospitalized); and Days 15 and 29 (if attends in-person visit or still hospitalized).
- Qualitative and quantitative PCR for SARS-CoV-2 in blood on Day 1; Days 3, 5, 8, and 11 (while hospitalized).
- Plasma proteomic analysis of cytokines and markers of inflammation including IL-17A, IL-22, and IL-1b on Days 1, 3, 8, 15, and 29 (if attends in-person visit or still hospitalized).
- Blood RNA transcriptome analysis on Days 1, 3, 8, 15, and 29 (if attends in-person visit or still hospitalized).
- PBMC assessment for phenotype and functional reactivity on Days 1, 3, 8, 15, and 29 (if attends in-person visit or still hospitalized; collected only at sites capable of collecting and processing PBMC).
- Serum samples for PK (at pre-dose, Day 5 (if hospitalized), Day 15, and Day 29) and serum samples for anti-drug antibodies and neutralizing antibodies at pre-dose and Day 29.

## 8.2 Safety and Other Assessments

Safety procedures and assessments are described in Section 8.2 of the Master protocol document. The total volume of blood collected over the course of this study for safety and research evaluations (including samples for secondary research-defined in master protocol section 10.1.1.2) is approximately 450 mL, with a maximum daily volume of approximately 73 mL.

#### 8.3 Adverse Events and Serious Adverse Events

AE reporting will occur as described in Section 8.3 of the Master protocol document.

#### 9. STATISTICAL CONSIDERATIONS

See Section 9 of Master protocol document.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

All supporting documentation and operational considerations are applicable to the entire platform trial and are not unique to the individual stages. These are therefore covered in the Master protocol document (Section 10).

#### 11. REFERENCES

- 1. Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, et al. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020:130(5):2620-9.
- 2. Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, et al. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020;395(10223):497-506.
- 3. Li G, Fan Y, Lai Y, Han T, Li Z, Zhou P, et al. Coronavirus infections and immune responses. J Med Virol. 2020;92(4):424-32.
- 4. Moore JB, June CH. Cytokine release syndrome in severe COVID-19. Science. 2020;368(6490):473-4.
- 5. Ye Q, Wang B, Mao J. The pathogenesis and treatment of the 'Cytokine Storm' in COVID-19. J Infect. 2020;80(6):607-13.
- 6. Hotez PJ, Bottazzi ME, Corry DB. The potential role of Th17 immune responses in coronavirus immunopathology and vaccine-induced immune enhancement. Microbes Infect. 2020;22(4-5):165-7.
- 7. Wu D, Yang XO. TH17 responses in cytokine storm of COVID-19: An emerging target of JAK2 inhibitor Fedratinib. J Microbiol Immunol Infect. 2020;53(3):368-70.
- 8. Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, et al. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020;8(4):420-2.
- 9. Faure E, Poissy J, Goffard A, Fournier C, Kipnis E, Titecat M, et al. Distinct immune response in two MERS-CoV-infected patients: can we go from bench to bedside? PLoS One. 2014;9(2):e88716.

- 10. Josset L, Menachery VD, Gralinski LE, Agnihothram S, Sova P, Carter VS, et al. Cell host response to infection with novel human coronavirus EMC predicts potential antivirals and important differences with SARS coronavirus. mBio. 2013;4(3):e00165-13.
- 11. Gaffen SL, Jain R, Garg AV, Cua DJ. The IL-23-IL-17 immune axis: from mechanisms to therapeutic testing. Nat Rev Immunol. 2014;14(9):585-600.
- 12. Toussirot E. The IL23/Th17 pathway as a therapeutic target in chronic inflammatory diseases. Inflamm Allergy Drug Targets. 2012;11(2):159-68.
- 13. SECURE-IBD database [Internet]. [cited 24 June 2020]. Available from: https://covidibd.org/.
- 14. Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, et al. Remdesivir for the Treatment of Covid-19 Preliminary Report. N Engl J Med. 2020.
- 15. U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (July 2017) 2017 [Available from:

https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf.